CLINICAL TRIAL: NCT04369170
Title: Changes on the Interproximal Marginal Bone Level After CAD-CAM Designed Bridges Directly Placed on Bone-level Implants, or With Intermediate Abutments. A Randomized Clinical Trial
Brief Title: Changes on the Interproximal Bone Level on Direct Prostheses or With Intermediate Abutments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Mozo Grau S.A. (Unknown)
Responsible Party: Principal Investigator, Juan Blanco Carrión, Professor, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ECIMG07/17
Record Dates: First submitted 2020-04-23; First posted 2020-04-30 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Periimplant Bone Loss; Marginal Periimplant Bone Level; Periimplantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: Parallel blinded clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participant and care provider are blinded, the outcomes assessor is also masked but the investigator knows if the participant belongs to group A or B when the data is recorded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A - Control Group (Other): Control group where an intermediate abutment is placed in between the CAD-CAM dental prostheses an the dental implant.
  Interventions: Device: Intermediate abutment
- Group B - Test Group (Experimental): Test group where the CAD-CAM dental prostheses is connected directly to the dental implant
  Interventions: Device: prosthesis connected directly to the implants

INTERVENTIONS:
Device: prosthesis connected directly to the implants — dental prostheses connected directly to the dental implants
  Arms: Group B - Test Group
Device: Intermediate abutment — dental prostheses connected with an intermediate abutment to the implant
  Arms: Group A - Control Group

SUMMARY:
Study Title: Changes on the Interproximal marginal bone level after CAD-CAM designed bridges directly placed on bone-level implants, or with intermediate abutments. A Randomized Clinical Trial.

* Objectives: To evaluate differences on changes on the interproximal marginal bone level 12 months after the connection of CAD/CAM designed prosthesis with an intermediate abutment (3mm long) or directly placed to bonelevel implants. Secondary objectives will be evaluate changes on the soft tissues and implant survival, as well as patients' satisfaction 3, 6 and 12 months after the connection of the definitive prosthesis.
* Design and Outcomes: Randomized double-blinded clinical trial with parallel design to asses the effect of CADCAM designed bridges directly placed
* Interventions and Duration: Patients will be selected according to the inclusion/exclusion criteria among those who attend the Unit of Periodontology of the University of Santiago de Compostela. After clinical and radiological implant planning, implant surgical placement will be scheduled. 2 MOZO GRAU® INHEX ST implants, with 3.75 mm or 4.25 mm of diameter and 8mm, 10mm or 11.5mm length will be placed on each patient, according to the bone availability. After 8 weeks of submerged healing, second stage surgery will be performed and definitive impression will be taken. All groups patients will keep a heeling abutment until the definitive prosthesis is placed, 3 weeks later (test group: direct to implant / control group: abutment 3 mm long). Clinical and radiological assessment after 1, 3, 6 and 12 months will be performed. Each participant will be on study about 15 months since the recruitment visit until the end of the study.
* Sample Size and Population: Based on previous studies, a sample size calculation determined that a group of 32 subjects, considering possible dropouts, will provide 80% power to detect a true radiographic difference of 0.80mm between groups after 12 months of observation since the definitive prosthesis connection. (Blanco et al 2017, Nóvoa et al 2017). A common standard deviation between groups was calculated (SD=0.715268015). A p ≤ 0.05 value will be considered significant (JM. Domenech & R. Granero 2010). A balanced random permuted block will be applied to prepare the randomization tables, stratifying for smoking habits (yes/no) with a 1:1 ratio between test and control groups.

DETAILED DESCRIPTION:
Changes on the interproximal periimplant marginal bone level measured as the distance between the bone crest to the first implant to bone contact, using periapical radiographs, will be evaluated.

Each patient will receive to implants that will be rehabilitated with an implant supported prosthesis, being the test group a prosthesis connected directly to the implants, while the control group will be a prosthesis connected to the implants through intermediate abutments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with systemic and periodontal health, over 18 years old, with a Plaque Index lower than 25%.

  * Patients with an absence of at least two contiguous teeth, with natural proximal teeth, excluding the anterior upper zone, allowing the rehabilitation with bridges with two implants and two to four prostheses units
  * Adequate bone quality available that allows the placement of MOZO GRAU® INHEX ST implants with diameters of 3.75 mm or 4.25 mm and lengths of 8, 10 and 11.5 mm.
  * At least 2mm of keratinized gingiva.
  * Natural antagonic teeth or implants with fixed restorations.

Exclusion Criteria:

* • Systemic Factors:

  * Long term use of systemic medication that may interfere with bone metabolism or medical conditions that require prolonged use of steroids and / or medication that may interfere with bone metabolism
  * History of leukocyte dysfunction and deficiency, immunodeficiency syndromes, renal failure or bonemetabolic disorders such as osteoporosis
  * Physical disabilities that may interfere with proper oral hygiene
  * Use of any medication or device in research for a period of 30 days prior to the implant surgery in the study
  * Alcoholism or drug abuse
  * Smoker of more than 10 cigarettes per day
  * Conditions or circumstances which could prevent compliance with the participation in the study or interfere with the analysis of the results, such as a history of non-compliance or lack of reliability.
  * Local Factors:
  * History of local radiotherapy
  * Bruxism
  * Mucosal diseases, such as Oral Lichen Planus
  * Not treated periodontitis
  * Persistent intraoral infection
  * Crestal bone regeneration less than 3 months before the implant placement
  * Not healed extraction sockets (less than 6 weeks post-extraction
  * Anterior aesthetic sextant of the maxilla

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2021-10-25 (Estimated); Study Completion 2022-10-25 (Estimated)

PRIMARY OUTCOMES:
Radiographic Periimplant Marginal Bone Loss | 12 months after the connection of the definitive prosthesis
  distance in millimetres measured on the periapical radiography between the implant neck and the first bone to implant contact after 12 months of loading

SECONDARY OUTCOMES:
Aesthetic parameters according to papilla refill between the prosthetic units | 12 months after the connection of the definitive prosthesis
  Using the Jemt index 1997 to evaluate the papilla refill between the prosthetic units
PROM's - Patient Recorded Outcomes Measurements | 12 months after the connection of the definitive prosthesis
  Visual Analogue Scale from 1 to 10 where the patient can evaluate the treatment according to aesthetics, chewing capacity, phonetics, confort and general satisfaction with the treatment
Adverse events | 12 months after the connection of the definitive prosthesis
  prostheses fracture, implant fracture, biological complications
probing pocket depth | 12 months after the connection of the definitive prosthesis
  measured with a CP12 calibrated periodontal probe from the gingival margin to the end of the periimplant pocket
Bleeding on probing | 12 months after the connection of the definitive prosthesis
  presence of bleeding after probing pocket depth using the Mombelli index 1987
Plaque index | 12 months after the connection of the definitive prosthesis
  presence of plaque on the implant supported rehabilitation using the Mombelli index 1987

CONTACTS AND LOCATIONS:
Locations (1):
- University of Santiago de Compostela, Santiago de Compostela, La Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alves CC, Munoz F, Cantalapiedra A, Ramos I, Neves M, Blanco J. Marginal bone and soft tissue behavior following platform switching abutment connection/disconnection--a dog model study. Clin Oral Implants Res. 2015 Sep;26(9):983-91. doi: 10.1111/clr.12385. Epub 2014 Apr 16. PMID 24735458
- [Background] Belser UC, Schmid B, Higginbottom F, Buser D. Outcome analysis of implant restorations located in the anterior maxilla: a review of the recent literature. Int J Oral Maxillofac Implants. 2004;19 Suppl:30-42. PMID 15635944
- [Background] Blanco J, Pico A, Caneiro L, Novoa L, Batalla P, Martin-Lancharro P. Effect of abutment height on interproximal implant bone level in the early healing: A randomized clinical trial. Clin Oral Implants Res. 2018 Jan;29(1):108-117. doi: 10.1111/clr.13108. Epub 2017 Dec 8. PMID 29222809
- [Background] Novoa L, Batalla P, Caneiro L, Pico A, Linares A, Blanco J. Influence of Abutment Height on Maintenance of Peri-implant Crestal Bone at Bone-Level Implants: A 3-Year Follow-up Study. Int J Periodontics Restorative Dent. 2017 Sep/Oct;37(5):721-727. doi: 10.11607/prd.2762. PMID 28817138
- [Background] Piao CM, Lee JE, Koak JY, Kim SK, Rhyu IC, Han CH, Herr Y, Heo SJ. Marginal bone loss around three different implant systems: radiographic evaluation after 1 year. J Oral Rehabil. 2009 Oct;36(10):748-54. doi: 10.1111/j.1365-2842.2009.01988.x. Epub 2009 Aug 20. PMID 19702681
- [Background] Tomasi C, Tessarolo F, Caola I, Wennstrom J, Nollo G, Berglundh T. Morphogenesis of peri-implant mucosa revisited: an experimental study in humans. Clin Oral Implants Res. 2014 Sep;25(9):997-1003. doi: 10.1111/clr.12223. Epub 2013 Jun 26. PMID 23799997